CLINICAL TRIAL: NCT05853406
Title: Determination of a Minimal Clinically Important Difference of the "Functional Reach Test" in the Elderly.
Status: Recruiting | Type: Observational
Sponsor: Pole Sante Grace de Dieu (Other)
Responsible Party: Sponsor
Other Study IDs: 20230102
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Functional Reach test — The determination by statistical research is carried out during a usual physiotherapy assessment of the volunteers. Data patient demographics and standard tests (FRT, Tinetti test, Timed Up and Go test, unipodal station) will be noted.
  A satisfaction questionnaire inspired by Patient rating of change will be sent to participants for the determination of the MCID by ANCHOR method.
  Concerning the Delphi method, a questionnaire will be sent to physiotherapists with proven geriatric activity.

SUMMARY:
The main objective of the study is to determine the Minimal Clinically Important Difference of the "Functional Reach Test" in the Elderly by a statistical method.

The first secondary objective of the study is to determine the Minimal Clinically Important Difference by the Anchor method based on a qualitative assessment by the patients of their own response. The second secondary objective is to determine the Minimal Clinically Important Difference by the Delphi method, based on the search for a consensus between physiotherapists specializing in geriatrics.

DETAILED DESCRIPTION:
The French population is aging, and geriatric rehabilitation care must adapt to this growing population. The functional reach test is a common clinical test in geriatrics. It helps to determine the risk of falling. However, its metrological qualities are not all determined. The Minimal Clinically Important Difference (MCID) is in particular unknown for this test. The MCID of a test makes it possible to personalize in a way more in-depth evaluation of physiotherapy treatment. So it is necessary to characterize this essential metrological determinant of a common balance skills assessment tool.

ELIGIBILITY:
Inclusion Criteria:

* People over 65 years old
* People in care with balance problems

Exclusion Criteria:

* People in an emergency situation
* People unable to give their consent (including people under guardianship)
* Patients already involved in another study.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The subjects recruited are patients aged over 65, having balance problems.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Functional Reach Test | 1 year
  Determination of MCID by statistical method

SECONDARY OUTCOMES:
Functional Reach Test | 1 year
  Determination of MCID by Patient rating of change
Functional Reach Test | 1 year
  Determination of MCID by Delphy Study

CONTACTS AND LOCATIONS:
Locations (1):
- PSLA GDD, Caen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosa MV, Perracini MR, Ricci NA. Usefulness, assessment and normative data of the Functional Reach Test in older adults: A systematic review and meta-analysis. Arch Gerontol Geriatr. 2019 Mar-Apr;81:149-170. doi: 10.1016/j.archger.2018.11.015. Epub 2018 Dec 7. PMID 30593986